CLINICAL TRIAL: NCT00653302
Title: Assessment of the Phenotype of the Type 2 Diabetic Responders to the First Insulinisation Using Lantus (Insulin Glargine) Plus Glucophage (Metformin) Combination After Failure in OADs Treatment
Brief Title: Phenotype Evaluation in Insulin Naive Patients Using Lantus (Insulin Glargine)
Acronym: GALATEE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Nathalie Billon/Study Director, sanofi-aventis France
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HOE901_4043
Record Dates: First submitted 2008-04-01; First posted 2008-04-04 (Estimated); Last update posted 2008-12-03 (Estimated); Status verified 2008-12

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine; Metformin

ARMS (1):
- 1 (Experimental): Lantus once a day plus Glucophage 1000mg, twice a day per os
  Interventions: Drug: Lantus (insulin glargine) + Glucophage (Metformin)

INTERVENTIONS:
Drug: Lantus (insulin glargine) + Glucophage (Metformin)

SUMMARY:
Primary objective:

* Efficacy assessment of the percentage of positive responders patients receiving Lantus plus glucophage association. Positive responders patients are defined by a final value of HbA1c<7% and/or a final decrease of HbA1c>15% compare to the basal value (HbA1c final - HbA1c basal).

Secondary objectives:

* Determination of the predictive criterion of HbA1c final,
* Determination of the predictive criterion of weight variation,
* Description of the glycemic and therapeutic criteria in the both groups of responders (positive and negative responders),
* Assessment of the lipidic parameters according to the HbA1c and weight changes during the study (final value - basal value).

Safety:

* Adverse Event (AE)/Serious Adverse Event (SAE) assessments

ELIGIBILITY:
Inclusion Criteria:

* Known type 2 diabetes for at least 2 years
* No history of Ketoacidosis
* BMI> 25 & <35 kg/m2
* Type 2 diabetes treated with oral bi or tritherapy for at least 6 months

  * With insulin release stimulator: sulfonamide or glinide at maximal posology (as defined in the SmPC),
  * and metformin at minimal posology 1700mg/day (1320 mg of metformin),
* HbA1c >= 7.5 and <11% for 2 different dosages during the last year

Exclusion Criteria:

* Type 1 diabetes
* Glucophage intolerability
* Pregnancy
* Breast feeding
* Partial pancreatectomy
* Hypersensitivity to insulin glargine excipient
* Renal failure with creatinin>135 µmol/L for male and >110 µmol/L for female patient
* Hepatitis with transaminases >3ULN
* Pre-proliferative or proliferative retinopathy
* Acute cardiovascular accident within the last 6 months
* Previous treatment with insulin within the last 6 months before randomization

Ages: 30 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2003-04; Primary Completion 2004-09 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
% of responders with HbA1c<7% and/or a final decrease of HbA1c>15% compare to the basal value (HbA1c final - HbA1c basal). | During the study conduct

SECONDARY OUTCOMES:
Determination of the predictive criterion of HbA1c final | During the study conduct
Determination of the predictive criterion of weight variation | During all the study conduct
HbA1c and weight variations (final value - basal value) | during the study
AE/SAE evaluation | from the informed consent signed up to the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Billon, Study Director — Sanofi-aventis administrative office France
Locations (1):
- Sanofi-aventis administrative office, Paris, France